CLINICAL TRIAL: NCT01441622
Title: In-hospital Assessment of the New Medical Device AL539 Developed for the Home Monitoring of Continuous Positive Airway Pressure (CPAP) Treatment in Patients With Obstructive Sleep Apnea Syndrome by Comparison With Respiratory Polygraphy
Brief Title: Evaluation of a New Medical Device AL539 in Patients With Obstructive Apneas Sleep Syndrome
Acronym: AL539
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Liquide Santé International (Industry)
Collaborators: Atlanstat (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ALMED-10-MD-030; IDR CB / 2010-A00923-36 (Other: AFSSAPS)
Record Dates: First submitted 2011-09-16; First posted 2011-09-27 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Continuous Positive Airway Pressure (CPAP); AL539; Home-monitoring
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AL539 (Experimental): Device AL539
  Interventions: Device: AL539 (SRETT)

INTERVENTIONS:
Device: AL539 (SRETT) — recording data with AL539 (SRETT)
  Other Names: Manufacturer name : SRETT

SUMMARY:
Continuous Positive Airway Pressure (CPAP) is the standard treatment in patients with Obstructive Sleep Apnea Syndrome (OSAS).

The goal of the study is to evaluate CPAP treatment duration recorded by the AL539 during attended in-hospital polysomnography in patients with Obstructive Sleep Apnea Syndrome.

DETAILED DESCRIPTION:
Patients are patients with sleep apnea predominantly obstructive, with CPAP for at least 2 months, and requiring in-hospital night polygraphic record control.

The medical device was developed to determine:

* the duration of use of CPAP by the patient,
* the persistence of any respiratory abnormalities during treatment.

These two parameters are used to ensure that treatment is done correctly.

The use of the AL539 is expected to improve the home-monitoring of ventilation with CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Sleep apnea predominantly obstructive
* CPAP for at least 2 months and requiring in-hospital night polygraphic record
* Written informed consent form
* Able to read and write in French

Exclusion Criteria:

* Ventilator with two levels of pressure
* CPAP breathing circuit non-compatible with the AL539
* Chronic respiratory disease
* Psychotropic treatment which may influence the respiratory parameters
* Acute rhinitis or acute nasopharyngitis
* Moderate or severe chronic heart failure
* CHEYNE-STOKES respiration
* Body mass index (BMI) > 40
* Pregnant woman or woman of childbearing potential with a positive urinary pregnancy test
* Uncontrolled progressive disease
* Psychiatric disorders or regular user of drugs
* Participation in any interventional clinical trial within 30 days prior to selection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
CPAP treatment duration | up to 12 hours
  Continous Positive Airway Pressure treatment duration

SECONDARY OUTCOMES:
Apneas-Hypopneas | up to 12 hours
  Apneas-Hypopneas Index (AHI) and Apneas Index (AI)
Mean pressure | up to 12 hours
  Mean pressure in patient circuit
Mean Flow | up to 12 hours
  Mean flow rate in patient circuit

CONTACTS AND LOCATIONS:
Overall Officials: Damien LEGER, Pr, Principal Investigator — Hôpital Hôtel Dieu
Locations (1):
- Hôpital Hôtel DIEU - Centre du sommeil et de la Vigilance, Paris, France

REFERENCES:
- [Derived] Leger D, Elbaz M, Piednoir B, Carron A, Texereau J. Evaluation of the add-on NOWAPI(R) medical device for remote monitoring of compliance to Continuous Positive Airway Pressure and treatment efficacy in obstructive sleep apnea. Biomed Eng Online. 2016 Feb 27;15:26. doi: 10.1186/s12938-016-0139-4. PMID 26922498